CLINICAL TRIAL: NCT03663244
Title: Is High Quality Effectiveness Research on Effective Stress Reduction in the Community Possible? -a Three-armed Parallel Pilot Trial in a Danish Municipality
Brief Title: Evaluating Effectiveness of Stress Reduction Programmes in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-03-3065
Record Dates: First submitted 2018-08-30; First posted 2018-09-10 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2018-08

CONDITIONS: Stress-related Problem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MindfulnessBasedStressReduction(MBSR) (Experimental): Standardised, curriculum-based MBSR-programme: 2.5-hour weekly group sessions over 8 weeks; one 6-hour silence retreat day; and 45 minutes daily homework 6 days a week.
  Interventions: Behavioral: MBSR
- Local Stress Reduction (LSR) (Experimental): Local stress reduction programme ; developed and delivered by two local psychologists. This programme is delivered in groups of 12 participants, in 2.5-hour weekly sessions over 8 weeks and includes approximately 10 minutes daily homework between the sessions.
  Interventions: Behavioral: LSR
- Wait-list (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: MBSR — Standardised stress reduction programme with established efficacy
  Arms: MindfulnessBasedStressReduction(MBSR)
Behavioral: LSR — Existing stress reduction programme in a Danish municipality
  Arms: Local Stress Reduction (LSR)

SUMMARY:
The aim was to assess the feasibility and to improve the quality of a definitive Randomised Controlled Trial (RCT) with the purpose to investigate the effectiveness of stress reduction programmes in the community. (A definitive RCT = an RCT with statistical power). Intermediate aims: to investigate 1) the potential generalizability: the accept among the target population (people with perceived stress) of participating in an RCT, including a description of the participant characteristics and the recruitment time ; 2) the risk of intervention effect dilution: the accept of allocated intervention in terms of programme completion ; 3) the risk of contamination: potential participation in (other) stress reduction treatment beyond the allocated intervention or non-intervention ; 4) the risk of selection problems or -bias: the lost to follow-up in the trial arms ; and finally, 5) the risk of information problems: the accept among participants of chosen outcome measurements, sensitivity of chosen outcome measures to detect effects, and indications of potential effects.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to understand, speak, and read Danish.

Exclusion Criteria:

* acute treatment-demanding clinical depression or a diagnosis of psychosis or schizophrenia
* abuse of alcohol, drugs, medicine
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Recruitment-rate | over 4 months
  Accept among total target group
Intervention-competition-rates participation | over 8 weeks
  Accept of the MBSR and the LSR programme defined by participation in >4 meetings
Proportions_other_treatment | over 8 weeks
  Risk of dilution of intervention effects. Proportions of allocated participants that have participated in other stress reduction treatment during the trial
Proportions_ lost-to-follow-up | over 8-10 weeks
  Risk of selection bias. Proportions of allocated participants lost to follow-up

SECONDARY OUTCOMES:
Proportions_Completed_PSS | twice over 8-10 weeks
  Proportions without missings in: Perceived Stress Scale
Proportions_Completed_SCL_5 | twice over 8-10 weeks
  Proportions without missings in: Symptom check list_5
Proportions_Completed_WHO_5 | twice over 8-10 weeks
  Proportions without missings in: WHO_5
Proportions_Completed_BRS | twice over 8-10 weeks
  Proportions without missings in: Brief Resiliens Scale
Proportions_Completed_ARSQ | twice over 8-10 weeks
  Proportions without missings in: Amsterdam Resting State Questionnaire
Proportions_Completed_FFMQ | twice over 8-10 weeks
  Proportions without missings in: Five Facet Mindfulness Questionnaire
Proportions_Completed_SCS | twice over 8-10 weeks
  Proportions without missings in: Neffs Self-Compassion-Scale
Proportions_Completed_EQ | twice over 8-10 weeks
  Proportions without missings in: Decentring scale
Proportions_measured_sysbp | twice over 8-10 weeks
  Proportions without missings in: systolic blood pressure
Proportions_measured_diabp | twice over 8-10 weeks
  Proportions without missings in: diastolic blood pressure
Proportions_measured_weight | twice over 8-10 weeks
  Proportions without missings in: weight
Proportions_measured_waist | twice over 8-10 weeks
  Proportions without missings in: waist
Proportions_completed_tova | twice over 8-10 weeks
  Proportions without missings in: TOVA-test
Proportions_measured_cholesterol | twice over 8-10 weeks
  Proportions without missings in: S-cholesterol
Proportions_measured_crp | twice over 8-10 weeks
  Proportions without missings in: C-Reaktivt Protein
Proportions_measured_il6 | twice over 8-10 weeks
  Proportions without missings in: inflammationmarker IL-6
Proposed_Effects_PSS | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_SCL_5 | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_WHO_5 | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_BRS | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects__ARSQ | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_FFMQ | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_SCS | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_EQ | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_sysbp | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_diabp | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_weight | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_waist | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_tova | over 8-10 weeks
  Differences between groups at 8-week follow
Proposed_Effects_cholesterol | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_crp | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
Proposed_Effects_il6 | over 8-10 weeks
  Differences with 95% Confidence intervals between groups at 8-week follow adjusted for baseline-value and adjusted for baseline-value, age, sex, educational level and history of mental disorder
dehydroepiandrosterone-sulfate (DHEAS) | over 8-10 weeks
  Plasma (µmol/L). Differences with 95% Confidence intervals between groups at 8-week follow

CONTACTS AND LOCATIONS:
Overall Officials: Lise Juul, PhD, Principal Investigator — Danish Center for Mindfulness, Department of Clinical Practice, Aarhus University
Locations (1):
- Aarhus University, Department of Clinical Medicine, Danish Center for Mindfulness, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juul L, Pallesen KJ, Bjerggaard M, Nielsen C, Fjorback LO. A pilot randomised trial comparing a mindfulness-based stress reduction course, a locally-developed stress reduction intervention and a waiting list control group in a real-life municipal health care setting. BMC Public Health. 2020 Mar 30;20(1):409. doi: 10.1186/s12889-020-08470-6. PMID 32228533